CLINICAL TRIAL: NCT03737851
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Assess the Safety and Efficacy of Elezanumab When Added to Standard of Care in Relapsing Forms of Multiple Sclerosis
Brief Title: A Study to Assess the Safety and Efficacy of Elezanumab When Added to Standard of Care in Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M18-918
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Relapsing multiple sclerosis; Multiple sclerosis; Elezanumab; ABT-555
MeSH Terms: conditions — Multiple Sclerosis | interventions — elezanumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to receive double-blind placebo by intravenous infusion.
  Interventions: Drug: placebo
- Elezanumab Dose 1 (Experimental): Participants randomized to receive double-blind elezanumab Dose 1 by intravenous infusion.
  Interventions: Drug: elezanumab
- Elezanumab Dose 2 (Experimental): Participants randomized to receive double-blind elezanumab Dose 2 by intravenous infusion.
  Interventions: Drug: elezanumab

INTERVENTIONS:
Drug: elezanumab — solution for infusion
  Other Names: ABT-555
  Arms: Elezanumab Dose 1; Elezanumab Dose 2
Drug: placebo — solution for infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of elezanumab in participants with relapsing Multiple Sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Participant has diagnosis of relapsing remitting multiple sclerosis (RRMS) or secondary-progressive multiple sclerosis (SPMS) with relapses within the past 24 months.
* Participant has cranial magnetic resonance imaging (MRI) demonstrating lesion(s) consistent with multiple sclerosis (MS).
* Participant has evidence of physical disability according to Expanded Disability Status Scale (EDSS) or Timed 25-Foot Walk (T25FW) or 9-Hole Peg Test.

Exclusion Criteria:

- Participants must not have experienced or be recovering from a clinical MS relapse within 6 months of Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (49):
- United States (42):
  - University of Alabama at Birmingham - Main /ID# 204618, Birmingham, Alabama
  - St. Josephs Hospital and Med Center /ID# 204197, Phoenix, Arizona
  - Sutter East Bay Medical Foundation-Jordon Research and Education Dev. Inst. /ID# 204249, Berkeley, California
  - The Research Center of Southern California /ID# 204269, Carlsbad, California
  - Vladimir Royter MD /ID# 204392, Hanford, California
  - UC Irvine Health /ID# 205728, Irvine, California
  - Stanford MS Center /ID# 204283, Palo Alto, California
  - UC Davis Health-Neurological Surgery /ID# 204188, Sacramento, California
  - UCSF School of Medicine - Neurology /ID# 204251, San Francisco, California
  - University of Colorado School of Medicine /ID# 204250, Aurora, Colorado
  - Advanced Neurosciences Research, LLC /ID# 204289, Fort Collins, Colorado
  - The University of Chicago Medical Center /ID# 205319, Chicago, Illinois
  - Indiana Univ School Medicine /ID# 204891, Indianapolis, Indiana
  - Rowe Neurology Institute /ID# 204391, Lenexa, Kansas
  - The NeuroMedical Center /ID# 204253, Baton Rouge, Louisiana
  - Ochsner Medical Center /ID# 204189, New Orleans, Louisiana
  - Duplicate_Parexel International /ID# 204273, Baltimore, Maryland
  - International Neurorehabilitation Institute /ID# 213332, Lutherville, Maryland
  - Pediatric Endocrine Associates /ID# 204279, Boston, Massachusetts
  - Michigan Institute for Neurological Disorders (MIND) /ID# 204194, Farmington Hills, Michigan
  - Memorial Neurological Institute and Center for Multiple Sclerosis /ID# 206328, Owosso, Michigan
  - Ridgeview Specialty Clinic Chaska - Neurology /ID# 204383, Chaska, Minnesota
  - Washington University-School of Medicine /ID# 204388, St Louis, Missouri
  - The MS Center for Innovations in Care at Missouri Baptist Medical Center /ID# 205433, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Cent /ID# 204745, Las Vegas, Nevada
  - Oklahoma Med Res. Foundation /ID# 204389, Oklahoma City, Oklahoma
  - Providence Neurological Specialties - West /ID# 204248, Portland, Oregon
  - Thomas Jefferson University /ID# 204281, Philadelphia, Pennsylvania
  - Advanced Neurosciences Institute /ID# 204557, Franklin, Tennessee
  - KCA Neurology - Franklin /ID# 204208, Franklin, Tennessee
  - Tri-State Mountain Neurology /ID# 204252, Johnson City, Tennessee
  - Neurology Consultants of Dallas - LBJ Fwy /ID# 204398, Dallas, Texas
  - UT HSC Multiple Sclerosis Research Group - Houston /ID# 206418, Houston, Texas
  - Dr. Bhupesh Dihenia, MD, PA /ID# 207839, Lubbock, Texas
  - Central Texas Neurology Consul /ID# 204268, Round Rock, Texas
  - Integrated Neurology Services, PLLC /ID# 204261, Alexandria, Virginia
  - Evergreen Neuroscience Institute /ID# 204203, Kirkland, Washington
  - Virginia Mason Medical Center /ID# 205440, Seattle, Washington
  - Swedish MS Center /ID# 204198, Seattle, Washington
  - University of Washington Medicine MS Center /ID# 205852, Seattle, Washington
  - West Virginia Univ School Med /ID# 204292, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital /ID# 204202, Milwaukee, Wisconsin
- Canada (7):
  - University of British Columbia - MS & NMO Clinical Trials Group, Djavad Mowafagh /ID# 204841, Vancouver, British Columbia
  - Duplicate_London Health Sciences Centre - University Hospital /ID# 204848, London, Ontario
  - Ottawa Hospital Research Institute /ID# 204842, Ottawa, Ontario
  - Unity Health Toronto - St. Michael's Hospital /ID# 206214, Toronto, Ontario
  - Recherche Sepmus Inc. /ID# 212851, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 204844, Montreal, Quebec
  - Montreal Neurological Institut /ID# 204843, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 208 subjects from 44 sites in the United States & Canada were enrolled into the study and were randomized: 208 subjects received at least 1 dose of study drug. Of the 208 subjects who received study drug, 182 completed treatment.
Period: Overall Study
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Started | 70 | 69 | 69
Completed | 62 | 63 | 57
Not Completed | 8 | 6 | 12

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) Analysis Set consists of all randomized subjects who received at least 1 dose of study drug. Subjects were grouped according to treatment as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2 | Total
Number analyzed (Participants) | 70 | 69 | 69 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 69 | 69 | 208
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 47 | 138
  Male | 24 | 24 | 22 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 6 | 20
  Not Hispanic or Latino | 60 | 65 | 63 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 60 | 62 | 62 | 184
  Non-White | 10 | 7 | 6 | 23
  Missing | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 5 | 4 | 10
  United States | 69 | 64 | 65 | 198
Type of Multiple Sclerosis (MS) [Count of Participants; unit: Participants]
  relapsing remitting MS (RRMS) | 66 | 67 | 66 | 199
  relapsing secondary-progressive MS (rSPMS) | 4 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Overall Response Score (ORS) at Week 52
Description: The ORS is a composite score derived from 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the non-dominant hand (9HPT-ND).
  Clinically significant worsening = -1, no change = 0, clinically significant improvement = +1.
  The ORS is the sum of these scores for the EDSS: Timed 25-Foot Walk, 9-Hole Peg Test-dominant, and 9-Hole Peg Test-nondominant and ranges from -4 to + 4.
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Number analyzed (Participants) | 59 | 61 | 55
score on a scale | 0.04 (0.175) | -0.17 (0.179) | -0.17 (0.177)

2. Secondary Outcome: Disability Improvement Response Rate
Description: Disability improvement response rate is assessed based on the Expanded Disability Status Scale Plus (EDSS+). EDSS+ is comprised of EDSS, Timed 25-Foot Walk (T25FW) and 9-Hole Peg Tests (9HPT).
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Number analyzed (Participants) | 70 | 69 | 69
Participants | 18 | 20 | 13
Statistical Analysis 1: Comparison: Placebo vs Elezanumab Dose 1; Logistic regression model for EDSS+ includes baseline values for EDSS, Timed 25-Foot Walk, 9-Hole Peg Test-dominant, 9-Hole Peg Test-nondominant, and treatment as a main effect. Subjects with missing values were imputed as non-responders; Test type: Other — a statistical test was not performed; Odds Ratio (OR) = 1.202, 95% CI 2-sided [0.559 to 2.584]
Statistical Analysis 2: Comparison: Placebo vs Elezanumab Dose 2; [analysis description as in outcome 2, analysis 1]; Test type: Other — a statistical test was not performed; Odds Ratio (OR) = 0.615, 95% CI 2-sided [0.266 to 1.421]

3. Secondary Outcome: Overall Response Score (ORS)
Description: The ORS is a composite score derived from 4 components: Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), 9-Hole Peg Test in the dominant hand (9HPT-D), and 9HPT in the non-dominant hand (9HPT-ND).
  Clinically significant worsening = -1, no change = 0, clinically significant improvement = +1.
  The ORS is the sum of these scores for the EDSS, Timed 25-Foot Walk, 9-Hole Peg Test-dominant and 9-Hole Peg Test-non-dominant and ranges from -4 to + 4.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Number analyzed (Participants) | 63 | 65 | 68
score on a scale | 0.05 (0.153) | -0.06 (0.159) | 0.12 (0.150)

4. Secondary Outcome: Overall Response Score (ORS)
Description: as for outcome 3
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Number analyzed (Participants) | 60 | 57 | 59
score on a scale | -0.04 (0.167) | -0.13 (0.175) | -0.06 (0.168)

5. Secondary Outcome: Overall Response Score (ORS)
Description: as for outcome 3
Time Frame: Week 36
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
Number analyzed (Participants) | 55 | 58 | 51
score on a scale | 0.09 (0.180) | -0.10 (0.184) | -0.17 (0.183)

ADVERSE EVENTS:
Time Frame: Up to 76 weeks
Description: Adverse Events were collected for all study participants, whether solicited or spontaneously reported by the study participant throughout the study, who received at least 1 dose of study drug and for a period of up to 39 weeks after the last dose of study drug.
Arm/Group | Placebo | Elezanumab Dose 1 | Elezanumab Dose 2
All-Cause Mortality (participants affected / at risk) | 1/70 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 6/70 | 7/69 | 4/69
Other Adverse Events (participants affected / at risk) | 52/70 | 48/69 | 54/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | Elezanumab Dose 1 (N=69) | Elezanumab Dose 2 (N=69)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL STRAIN (Investigations) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
UHTHOFF'S PHENOMENON (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | Elezanumab Dose 1 (N=69) | Elezanumab Dose 2 (N=69)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 5 (5) | 6 (6)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 3 (3) | 6 (6)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
FATIGUE (General disorders) | 10 (16) | 4 (4) | 8 (10)
PAIN (General disorders) | 5 (5) | 1 (1) | 3 (4)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3) | 6 (6)
INFLUENZA (Infections and infestations) | 2 (2) | 3 (3) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 5 (5) | 5 (5)
SINUSITIS (Infections and infestations) | 3 (4) | 2 (2) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 6 (7)
URINARY TRACT INFECTION (Infections and infestations) | 10 (19) | 9 (15) | 10 (12)
FALL (Injury, poisoning and procedural complications) | 12 (14) | 11 (16) | 10 (13)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 6 (23) | 5 (9) | 6 (12)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 3 (3) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (9) | 4 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 4 (4)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 2 (3)
DIZZINESS (Nervous system disorders) | 3 (3) | 3 (5) | 4 (5)
HEADACHE (Nervous system disorders) | 8 (13) | 9 (13) | 5 (6)
MIGRAINE (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 5 (6) | 6 (8) | 6 (6)
MUSCLE SPASTICITY (Nervous system disorders) | 1 (1) | 5 (5) | 5 (5)
ANXIETY (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4)
INSOMNIA (Psychiatric disorders) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT03737851/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03737851/SAP_001.pdf